CLINICAL TRIAL: NCT04090125
Title: Improving Physical Activity and Gait Symmetry After Total Knee Arthroplasty
Acronym: PAS-TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-0568; R21AR074149-01A1 (NIH)
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2022-12

CONDITIONS: Knee Replacement, Total; Knee Arthroplasty, Total
Keywords: knee; total knee replacement; physical therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity and Symmetry (PAS) Intervention (Experimental): Participants assigned to the PAS intervention will receive 4 sessions on balance training and physical activity coaching delivered by a physical therapist, in addition to their usual post-TKA physical therapy (PT) care.
  Interventions: Behavioral: PAS Intervention
- Attention Control (Placebo Comparator): Participants assigned to the ATT group will receive usual post-TKA physical therapy (PT) care, followed by two additional sessions with their physical therapist.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: PAS Intervention — The PAS program will be initiated during the final usual care PT visits. The PAS content will be included within the last two routine PT visits (Sessions 1 and 2). Session 1 will emphasize the importance of PA in TKA recovery, work with participants to establish SMART goals regarding overall PA and provide community-based and other resources to support overall PA. Session 2 will include balance exercise content to improve joint loading symmetry and home exercises will be assigned. Then, PAS participants will receive a follow-up phone call after 4 weeks (to assist with activity progression and problem-solving) and an additional in-person visit after 8 weeks (to visually monitor exercise performance and re-assess proportional weight-bearing ability).
  Arms: Physical Activity and Symmetry (PAS) Intervention
Behavioral: Attention Control — This will include usual in-person post TKA PT followed by 2 additional contacts (Session 1 and 2) with the physical therapist. Session 1 (phone) will review recovery benchmarks, assessment of participants' daily activities and reminders about symptoms that should trigger contacting a medical professional. Session 2 (in-person) will involve physical performance tests and comparison to appropriate normative values.
  Arms: Attention Control

SUMMARY:
The purpose of this pilot study is to examine the effectiveness of the Physical Activity and Symmetry (PAS) program, compared to an attention (ATT)control group, for patients with post-total knee arthroplasty (TKA). The investigators hypothesize that the PAS treatment will result in meaningful improvements in physical activity (PA) and joint loading symmetry compared to the ATT group.

DETAILED DESCRIPTION:
Background and Significance: Total knee arthroplasty (TKA) has been shown to decrease pain and to improve range of motion and some aspects of physical function. However, accumulating evidence shows that patients have persistent deficits in other critical outcomes following TKA. First, the majority of patients do not substantially increase physical activity beyond levels prior to TKA, remaining well below Department of Health and Human Services recommendations and levels of healthy individuals. This has serious negative implications for both joint health and overall health. Second, studies show that gait asymmetries are common following TKA, such that patients continue to load the non-surgical leg more heavily during walking, even when the post-surgical leg is pain free. This places the contralateral limb at risk for developing or worsening osteoarthritis. Other research shows there is large variability in post-TKA rehabilitation, along with sub-optimal exercise content. Collectively, these findings emphasize the critical need to improve the post-TKA rehabilitation process. However, there are currently no evidence-based approaches to improve overall physical activity and deficits in joint loading symmetry that have been identified following TKA.

Study Aims: This research project will provide important preliminary information on the novel post-TKA PAS program through achieving the following specific aims: 1) Obtain preliminary data on the efficacy of the PAS program with respect to the change in objectively assessed physical activity, measured via accelerometers; 2) Obtain preliminary data on the efficacy of the PAS program with respect to change in peak load symmetry during walking, measured by a novel 3-sensor insole device; 3) Assess the feasibility and acceptability of the PAS program following TKA.

Study Description: Investigators will conduct an exploratory randomized controlled study, with n=60 patients >=18 years receiving post-TKA physical therapy (PT) at a UNC Healthcare System clinic. Patients will be equally allocated to the PAS intervention or an attention (ATT) control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving post-total knee arthroplasty (TKA) physical therapy (PT) at a University of North Carolina (UNC) Healthcare System clinic

Exclusion Criteria:

* significant cognitive impairment
* neurological disorders affecting gait
* systemic rheumatic disease
* hospitalization for a cardiovascular condition the past six months
* psychosis
* substance abuse disorder
* lower extremity surgery in the past year
* any other health conditions determined to be contraindications to a home exercise program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2023-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli D Allen, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Thurston Arthritis Research Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: SAP
Time Frame: Data will become available following publication of primary and secondary outcomes, and data will be available until the study is closed with the local IRB.
Access Criteria: Data will be accessible following publication of study results and will be available until the study is closed with the local IRB.

RESULTS

PARTICIPANT FLOW:
Groups:
- Attention Control: Participants assigned to the Attention Control (ATT) group will receive usual post-TKA physical therapy (PT) care, followed by two additional sessions with their physical therapist.
  Attention Control: This will include usual in-person post TKA PT followed by 2 additional contacts (Session 1 and 2) with the physical therapist. Session 1 (phone) will review recovery benchmarks, assessment of participants' daily activities and reminders about symptoms that should trigger contacting a medical professional. Session 2 (in-person) will involve physical performance tests and comparison to appropriate normative values.
Period: Overall Study
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Started | 30 | 30
Completed 3-month Follow-up | 23 | 24
Completed (Completed 6-month follow-up assessment) | 20 | 24
Not Completed | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (7.8) | 66.1 (7.2) | 66.2 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 30 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 23 | 23 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 3 in Objectively Assessed Physical Activity (Accelerometer)
Description: Minutes of moderate to vigorous intensity PA (MVPA) per week measured via accelerometer.
  A log transformation was applied due to superior diagnostics relative to untransformed values in statistical modeling; transformed values are presented here.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: Minutes per week
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 23 | 24
Minutes per week | 0.59 [0.12 to 1.07] | 0.36 [-0.12 to 0.84]
Statistical Analysis 1: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Test type: Superiority; p = 0.485, Mixed Models Analysis; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.90 to 0.43]

2. Primary Outcome: Change From Baseline to Month 6 in Objectively Assessed Physical Activity (Accelerometer)
Description: as for outcome 1
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: Minutes per week
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 20 | 24
Minutes per week | 0.12 [-0.34 to 0.57] | 0.64 [0.23 to 1.06]
Statistical Analysis 1: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Test type: Superiority; p = 0.0887, Mixed Models Analysis; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-1.13 to 0.08]

3. Primary Outcome: Change From Baseline to Month 3 in Peak Joint Load Symmetry During Walking
Description: Participants will complete a 10 meter walking test while load beneath each foot is recorded using an instrumented insole. Loading symmetry (peak ground reaction force) will be assessed using the limb symmetry index (LSI (|Surgical/Non-Surgical|*100), values lower than 100% indicate less loading of the surgical limb.
  A log transformation was applied due to superior diagnostics relative to untransformed values in statistical modeling; transformed values are presented here.
Time Frame: Baseline, Month 3
Population: This includes all participants with available insole data at baseline and 6-month follow-up. Some participants did not have usable insole data due to technical issues
Measure: Mean (95% Confidence Interval); unit: percentage of non-surgical limb force
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 15 | 19
percentage of non-surgical limb force | 0.04 [-0.04 to 0.13] | -0.02 [-0.09 to 0.06]
Statistical Analysis 1: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Test type: Superiority; p = 0.296, Mixed Models Analysis; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.05 to 0.13]

4. Primary Outcome: Change From Baseline to Month 6 in Peak Joint Load Symmetry During Walking
Description: as for outcome 3
Time Frame: Baseline, Month 6
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: percentage of non-surgical limb force
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 13 | 18
percentage of non-surgical limb force | -0.05 [-0.11 to 0.01] | 0.02 [-0.03 to 0.07]
Statistical Analysis 1: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Test type: Superiority; p = 0.094, Mixed Models Analysis; Mean Difference (Final Values) = -0.07, 95% CI 2-sided [-0.15 to 0.01]

5. Secondary Outcome: Change From Baseline to Month 3 in Self-Reported Physical Activity.
Description: Self-Reported Physical Activity will be assessed using the Modified version of the CHAMPS (Community Health Activities Model Program for Seniors) Physical Activity Measure. Data from the questionnaire is used to determine variety, frequency, and minutes per week from physical activity. This outcome pertains to minutes of physical activity of moderate or greater intensity (metabolic equivalents ≥ 3.0). A square root transformation was applied due to superior diagnostics relative to untransformed values in statistical modeling; transformed values are presented here.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: minutes per week
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 23 | 24
minutes per week | 3.23 [-0.24 to 6.71] | -0.62 [-4.02 to 2.77]
Statistical Analysis 1: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Test type: Superiority; p = 0.11, Mixed Models Analysis; Mean Difference (Final Values) = 3.85, 95% CI 2-sided [-0.91 to 8.62]

6. Secondary Outcome: Change From Baseline Month 6 in Self-Reported Physical Activity.
Description: as for outcome 5
Time Frame: Baseline to Month 6
Measure: Mean (95% Confidence Interval); unit: Minutes per week
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 20 | 24
Minutes per week | 1.58 [-2.71 to 5.87] | -0.16 [-4.23 to 3.90]
Statistical Analysis 1: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Test type: Superiority; p = 0.55, Mixed Models Analysis; Mean Difference (Final Values) = 1.74, 95% CI 2-sided [-4.10 to 7.59]

7. Secondary Outcome: Change From Baseline to Month 3 in Steps Per Day
Description: Step counts measured via accelerometer. A log transformation was applied due to superior diagnostics relative to untransformed values in statistical modeling; transformed values are presented here.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: steps per day
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 23 | 24
steps per day | 0.18 [0.04 to 0.32] | 0.33 [0.19 to 0.46]
Statistical Analysis 1: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Test type: Superiority; p = 0.134, Mixed Models Analysis; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.34 to 0.05]

8. Secondary Outcome: Change From Baseline to Month 6 in Steps Per Day
Description: as for outcome 7
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: steps per day
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 20 | 24
steps per day | 0.15 [-0.01 to 0.30] | 0.32 [0.18 to 0.46]
Statistical Analysis 1: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Test type: Superiority; p = 0.09, Mixed Models Analysis; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.38 to 0.03]

9. Secondary Outcome: Change From Baseline to Month 3 in Minutes of Any Physical Activity (PA)
Description: Minutes of any PA measured via accelerometer. A log transformation was applied due to superior diagnostics relative to untransformed values in statistical modeling; transformed values are presented here.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 23 | 24
minutes per day | 0.04 [-0.04 to 0.11] | 0.09 [0.02 to 0.17]
Statistical Analysis 1: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Test type: Superiority; p = 0.25, Mixed Models Analysis; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.16 to 0.04]

10. Secondary Outcome: Change From Baseline to Month 6 in Minutes of Any Physical Activity (PA)
Description: as for outcome 9
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 20 | 24
minutes per day | 0.00 [-0.01 to 0.01] | 0.09 [0.00 to 0.18]
Statistical Analysis 1: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Test type: Superiority; p = 0.16, Mixed Models Analysis; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.22 to 0.04]

11. Secondary Outcome: Change From Baseline to Month 3 in Sedentary Minutes
Description: Minutes of sedentary activity per day, measured via accelerometer
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: minutes per day
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 23 | 24
minutes per day | -5.32 [-27.52 to 16.89] | -26.68 [-48.70 to -4.65]
Statistical Analysis 1: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Test type: Superiority; p = 0.167, Mixed Models Analysis; Mean Difference (Final Values) = 21.36, 95% CI 2-sided [-9.29 to 52.02]

12. Secondary Outcome: Change From Baseline to Month 6 in Sedentary Minutes
Description: Minutes of sedentary activity per day, measured via accelerometer
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 23 | 24
minutes | -1.37 [-29.66 to 26.92] | -26.52 [-52.47 to -0.56]
Statistical Analysis 1: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Test type: Superiority; p = 0.189, Mixed Models Analysis; Mean Difference (Final Values) = 25.15, 95% CI 2-sided [-12.85 to 63.14]

13. Secondary Outcome: Change From Baseline to Month 3 in Berg Balance Scale
Description: Berg Balance Scale includes 14 tests of static and dynamic balance. Each item is scored along a 5-point scale, ranging from 0 to 4. Zero indicates the lowest level of function and 4 the highest level of function. The total score ranges from 0 to 56. Lower scores indicate reduced functional mobility.
Time Frame: Baseline, Month 3
Population: We had to discontinue administration of balance measures for this study for an extended period of time due to COVID-19, as these tests require the test administrator to be in close proximity to the person being tested. Only 1 person completed all components of this balance test at both baseline and 3-month follow-up.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 0 | 1
score on a scale |  | -4 [-4 to -4]

14. Secondary Outcome: Change From Baseline to Month 6 in Berg Balance Scale
Description: as for outcome 13
Time Frame: Baseline, Month 6
Population: We had to discontinue administration of balance measures for this study for an extended period of time due to COVID-19, as these tests require the test administrator to be in close proximity to the person being tested. No participants completed all components of this balance test at both baseline and 6-month follow-up.
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Change From Baseline to Month 3 in Brief Balance Evaluation Systems Test
Description: Brief Balance Evaluation Systems includes 8 tasks across 6 domains. Each item is scored: 0-3 points (0 representing severe impairment and 3 representing no balance impairment), score range is 0-24). Lower scores indicate higher levels of balance impairment.
Time Frame: Baseline, Month 3
Population: as for outcome 13
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 0 | 1
score on a scale |  | 1 [1 to 1]

16. Secondary Outcome: Change From Baseline to Month 6 in Brief Balance Evaluation Systems Test
Description: Brief Balance Evaluation Systems includes 8 tasks across 6 domains. Each item is scored: 0-3 points (0 representing severe impairment and 3 representing no balance impairment), score range is 0-24. Lower scores indicate higher levels of balance impairment.
Time Frame: Baseline, Month 6
Population: as for outcome 14
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Change From Baseline to Month 3 in Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: The KOOS is a patient-reported outcome measurement instrument, developed to assess the patient's opinion about their knee and associated problems. Five KOOS subscale scores were administered: Pain (9 items), Symptoms (7 items), Function in daily living (17 items), Function in Sport and Recreation (5 items), and knee-related Quality of Life (4 items). All items are scored on 5-point Likert scales. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Time Frame: Baseline, Month 3
Population: Only 1 participant answered enough questions on the Function and Sport and Recreation Subscale to score this subscale, per instrument instructions. This is because in this post-surgical sample many still had activity restrictions and had been instructed to not yet engage in many of the activities on this subscale.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 23 | 24
score on a scale
  Pain | 28.70 [24.24 to 33.16] | 26.19 [21.80 to 30.58]
  Symptoms | 23.16 [17.76 to 28.56] | 22.02 [16.72 to 27.32]
  Quality of Life | 29.12 [22.08 to 36.16] | 32.66 [25.77 to 39.54]
  Function in Daily Living | 20.91 [17.90 to 23.92] | 18.37 [15.41 to 21.33]
  Function in Sport and Recreation: number analyzed (Participants) | 1 | 1
  Function in Sport and Recreation | 41.7 | 0
Statistical Analysis 1: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Pain subscale; Test type: Superiority; p = 0.42, Mixed Models Analysis; Mean Difference (Final Values) = 2.51, 95% CI 2-sided [-3.65 to 8.67]
Statistical Analysis 2: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Symptoms subscale; Test type: Superiority; p = 0.76, Mixed Models Analysis; Mean Difference (Final Values) = 1.14, 95% CI 2-sided [-6.29 to 8.57]
Statistical Analysis 3: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Quality of life subscale; Test type: Superiority; p = 0.46, Mixed Models Analysis; Mean Difference (Final Values) = -3.54, 95% CI 2-sided [-13.20 to 6.12]
Statistical Analysis 4: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Function in daily life; Test type: Superiority; p = 0.22, Mixed Models Analysis; Mean Difference (Final Values) = 2.54, 95% CI 2-sided [-1.61 to 6.69]

18. Secondary Outcome: Change From Baseline to Month 6 in Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: The KOOS is a patient-reported outcome measurement instrument, developed to assess the patient's opinion about their knee and associated problems. Five KOOS subscale scores were administered: Pain (9 items), Symptoms (7 it4ems) Function in daily living (17 items), Function in Sport and Recreation (5 items), and knee-related Quality of Life (4 items). All items are scored on 5-point Likert scales. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Time Frame: Baseline, Month 6
Population: Only 2 participants answered enough questions on the Function and Sport and Recreation Subscale to score this subscale, per instrument instructions. This is because in this post-surgical sample many still had activity restrictions and had been instructed to not yet engage in many of the activities on this subscale. Therefore only four of the subscales were scored and analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 20 | 24
score on a scale
  Pain | 30.16 [25.43 to 34.89] | 28.72 [24.26 to 33.19]
  Symptoms | 29.49 [23.67 to 35.31] | 25.54 [20.04 to 31.04]
  Quality of life | 36.47 [28.13 to 44.80] | 34.83 [27.05 to 42.61]
  Function in daily life | 22.92 [19.26 to 26.57] | 19.67 [16.29 to 23.04]
  Function in Sport and Recreation: number analyzed (Participants) | 1 | 1
  Function in Sport and Recreation | 22.9 | 41.7
Statistical Analysis 1: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Pain subscale; Test type: Superiority; p = 0.65, Mixed Models Analysis; Mean Difference (Final Values) = 1.43, 95% CI 2-sided [-4.98 to 7.85]
Statistical Analysis 2: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Symptoms subscale; Test type: Superiority; p = 0.32, Mixed Models Analysis; Mean Difference (Final Values) = 3.95, 95% CI 2-sided [-3.93 to 11.83]
Statistical Analysis 3: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Quality of life; Test type: Superiority; p = 0.77, Mixed Models Analysis; Mean Difference (Final Values) = 1.64, 95% CI 2-sided [-9.61 to 12.89]
Statistical Analysis 4: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Function in daily life; Test type: Superiority; p = 0.19, Mixed Models Analysis; Mean Difference (Final Values) = 3.25, 95% CI 2-sided [-1.67 to 8.17]

19. Secondary Outcome: Change From Baseline to Month 3 in Tampa Scale for Kinesiophobia
Description: The Tampa Scale of Kinesiophobia is a 17 item scale for assessing fear of movement. The scale specifically assesses activity avoidance due to pain-related fear of movement. All items are measured on a 4-point scale from "strongly agree" to "strongly disagree." A score of 17 is the lowest possible score, and indicates no kinesiophobia or negligible. A score of 68 is the highest possible score and indicates extreme fear of pain with movement.
Time Frame: Baseline, Month 3
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 23 | 24
units on a scale | -4.81 [-6.98 to -2.65] | -2.86 [-4.94 to -0.78]
Statistical Analysis 1: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Test type: Superiority; p = 0.191, Mixed Models Analysis; Mean Difference (Final Values) = -1.95, 95% CI 2-sided [-4.92 to 1.01]

20. Secondary Outcome: Change From Baseline to Month 6 in Tampa Scale for Kinesiophobia
Description: as for outcome 19
Time Frame: Baseline, Month 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
Number analyzed (Participants) | 20 | 24
units on a scale | -8.31 [-10.41 to -6.20] | -2.86 [-4.81 to -0.90]
Statistical Analysis 1: Comparison: Physical Activity and Symmetry (PAS) Intervention vs Attention Control; Test type: Superiority; p = 0.0004, Mixed Models Analysis; Mean Difference (Final Values) = -5.45, 95% CI 2-sided [-8.28 to -2.62]

ADVERSE EVENTS:
Time Frame: Approximately 6 months for each participant (enrollment to completion of 6-month follow-up assessment)
Arm/Group | Physical Activity and Symmetry (PAS) Intervention | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 6/30 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Activity and Symmetry (PAS) Intervention (N=30) | Attention Control (N=30)
Distal radius fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — fall while walking on uneven pavement, resulting in left intra-articular distal radius fracture; treated with open reduction and internal fixation
Heart palpitations (Cardiac disorders) | 1 (1) | 0 (0) — Participants presented at emergency department, assessments conducted, all markers normal, not admitted
Senile nuclear sclerosis, bilateral (Eye disorders) | 1 (1) | 0 (0) — Resolved with treatment
Cystitis (Infections and infestations) | 1 (1) | 0 (0) — Patient present to emergency department (ED) for evaluation of urinary changes. Not admitted.
Fatigue, shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient presented to ED with c/o shortness of breath (SOB), fatigue; Computed Tomography (CT) scan did not show any pulmonary embolism or blood clots, did not show anything wrong with the heart or lungs, pt not admitted
Postoperative pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient struggled postoperative pain relief; plans were made for manipulation of the left knee under anesthesia, discharged same day
Cataract surgery (Eye disorders) | 1 (1) | 0 (0) — discharged same day

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT04090125/Prot_001.pdf
  • Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT04090125/SAP_002.pdf
  • Informed Consent Form (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT04090125/ICF_003.pdf